CLINICAL TRIAL: NCT01536171
Title: Peak Impact Forces and Metabolic Cost During Mid-Forefoot Striking in Shod Versus Barefoot Runners: A Pilot Study
Brief Title: Peak Impact Forces and Metabolic Cost During Mid-Forefoot Striking in Shod Versus Barefoot Runners
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 497-2010
Record Dates: First submitted 2011-11-02; First posted 2012-02-20 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: runners; mid-foot strike; fore foot strike; metabolic costs; trained runners (men,women) with a FM strike; shod running; barefoot running
MeSH Terms: interventions — Running

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Shod versus Barefoot Running: two running conditions, with normal running shoes and barefoot
  Interventions: Other: running with normal running shoes and barefoot

INTERVENTIONS:
Other: running with normal running shoes and barefoot — shod condition: normal running shoes barefoot condition: running with no shoewear

SUMMARY:
This experimental study will compare impact forces and metabolic cost in runners (N=20; ages 18-45 years, who already use a forefoot strike running gait) in two treadmill running test sessions (shod vs barefoot running)

DETAILED DESCRIPTION:
Specific Aim 1: To identify if differences in metabolic cost exist between barefoot versus cushioned shod FM strikers during an acute bout of running exercise. Hypothesis: The metabolic cost will be higher in the cushioned shod runners with forefoot and midfoot strike compared to the barefoot runners.

Specific Aim 2: To identify if differences in peak impact forces exist between barefoot versus cushioned shod runners in forefoot-midfoot (FM) strikers.

Hypothesis: Peak impact forces will be higher in the barefoot runners with a forefoot and midfoot striking running style compared to the cushioned shod runners with a forefoot and midfoot striking running style.

ELIGIBILITY:
Inclusion Criteria:

* trained runners with a running foot striking style of either initial forefoot or midfoot strike.
* run on average at least 20 miles/week
* be able to run for at least 20 minutes at one session
* free of any orthopedic limitation

Exclusion Criteria:

* history of lower extremity injury within the last 6 months prior to testing
* rear-foot strike running style
* does not run in a cushioned shoe on any occasion
* runs on average < 20 miles/week
* unable to run for 20 minutes or greater
* presence of any open wound or deformity on the feet which would prevent participant from running barefoot
* neurologic injury that would preclude normal running activity.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: trained runners (men and women) who run with a FM strike (self-reported and verified in the laboratory).
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather K Vincent, PhD, Principal Investigator — University of Florida
Locations (1):
- UF&Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mid-Forefoot Striking in Shod Versus Barefoot Runners: trained runners (men,women) with a FM strike (verified in the lab)
Period: Overall Study
Arm/Group | Mid-Forefoot Striking in Shod Versus Barefoot Runners
Started | 22
Completed | 21
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Healthy young active adults
Arm/Group | Mid-Forefoot Striking in Shod Versus Barefoot Runners
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Secondary Outcome: Peak Impact Forces During Barefoot and Shod Running
Description: This study will be measuring the peak impact forces that a runner produces when running on the treadmill with shoes (shod) and without shoes.
  Each person will run for 20 minutes on the treadmill on two different days, one with and one day without shoes.
Time Frame: Study consists of two visits, approximately 2 hours for each visit
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | Mid-Forefoot Striking in Shod Versus Barefoot Runners
Number analyzed (Participants) | 22
Newtons
  Peak Impact forces during shod running | 1756 (310)
  Peak impact during barefoot running | 1703 (285)

2. Primary Outcome: Metabolic Rate During Barefoot and Shod Running
Description: This study will measure the metabolic rate when a person runs on the treadmill with shoes (shod) and without shoes.
  Each person will run for 20 minutes on the treadmill on two different days, one with and one day without shoes.
Time Frame: Study consists of two visits, approximately 2 hours for each visit
Measure: Mean (Standard Deviation); unit: kilojoules per minute
Groups:
- Mid-Forefoot Striking in Shod Versus Barefoot Runners: two running conditions, with normal running shoes and barefoot
Arm/Group | Mid-Forefoot Striking in Shod Versus Barefoot Runners
Number analyzed (Participants) | 22
kilojoules per minute
  Metabolic rate shod running | 57.8 (7.8)
  Metabolic rate barefoot running | 57.5 (8.4)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Mid-Forefoot Striking in Shod Versus Barefoot Runners
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 1/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mid-Forefoot Striking in Shod Versus Barefoot Runners (N=22)
irritation to bottom of foot when running barefoot (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No